CLINICAL TRIAL: NCT06524440
Title: Comorbidities and the Management of Hypertensive Heart Disease in a Low-Resource Setting: A Cross-Sectional Study
Brief Title: Hypertensive Heart Disease in DR Congo
Status: Recruiting | Type: Observational
Sponsor: Association of Future African Neurosurgeons, Yaounde, Cameroon (Other)
Responsible Party: Sponsor
Other Study IDs: AAfricanNeuro
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Hypertensive Heart Disease
Keywords: Comorbidities; Democratic Republic of Congo; Hypertensive heart disease; Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this Cross-sectional study, we will analyzed data from a tertiary referral Congolese hospital to find whether or not Congolese patients with hypertensive heart disease have multiple comorbid conditions. Will report on the management and outcomes of the patients.

DETAILED DESCRIPTION:
This will be done by collecting individual data on BMI, dyslipidemia, stroke, diabetes, serum creatinine, HDL, LDL, and urea levels for patients diagnosed with hypertensive heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients is 18 year or older
* Patient is diagnosed with hypertensive heart disease

Exclusion Criteria:

* Patient is not 18 year or older
* Patient is not diagnosed with hypertensive heart disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients 18 year or older diagnosed with hypertensive heart disease at Monkole Mother and Infant Hospital Center from January to December 2019
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-07-26 (Estimated); Primary Completion 2024-07-28 (Estimated); Study Completion 2024-07-29 (Estimated)

PRIMARY OUTCOMES:
High Systolic Blood Pressure | 1 month
  The study will use high systolic blood pressures as a measure for hypertensive heart disease.

CONTACTS AND LOCATIONS:
Overall Officials: Raïssa K Kongue, MD, Principal Investigator — Faculty of Medicine, Bel Campus University of Technology, Kinshasa, Democratic Republic of Congo
Locations (1):
- Monkole Mother and Infant Hospital Center, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
The IPD from this study will be openly available in the Open Science Framework.
Time Frame: It will be indefinitely available after the study has been conducted.
Access Criteria: This data will be open to all individuals.
URL: http://osf.io